CLINICAL TRIAL: NCT06483451
Title: Hepatitis C Virus Management Through Facilitated Telemedicine Integrated Into Opioid Treatment Programs: Catholic Health System Experience
Brief Title: Facilitated Telemedicine in the Catholic Health System
Status: Not yet recruiting | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Andrew Talal, Professor of Medicine, State University of New York at Buffalo
Other Study IDs: STUDY00008372
Record Dates: First submitted 2024-06-14; First posted 2024-07-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: HCV
Keywords: telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals with active HCV infection: Individuals with active HCV infection

SUMMARY:
Hepatitis C virus is a leading cause of morbidity and mortality globally with the highest prevalence and incidence among people with opioid use disorder. We aim to establish facilitated telemedicine as a standard of care treatment approach at 3 opioid treatment programs operated by the Catholic Health System. This study is a chart review data analysis to evaluate outcomes of facilitated telemedicine integrated into opioid treatment programs and to evaluate the number of individuals who initiate and complete treatment for hepatitis C virus infection.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) is a leading cause of morbidity and mortality globally with the highest prevalence and incidence among people with opioid use disorder. In 2013, direct-acting antivirals were introduced for HCV treatment: all oral medications with minimal side effects and excellent efficacy when taken for 2-3 months. However, only 34% of eligible individuals received direct-acting antivirals between 2013 and 2022. Moreover, HCV treatment with direct-acting antivirals was substantially lower among people with opioid use disorder. Access to highly effective HCV treatment by the populations with the greatest need remains inadequate.

To address this issue, we propose that facilitated telemedicine could be a bridge to integrate HCV treatment into opioid treatment programs. In our model, telemedicine encounters are facilitated by a case manager who is also a patient advocate and an educator. We recently completed a randomized clinical trial that compared facilitated telemedicine integrated into opioid treatment programs for HCV treatment compared to offsite referral. The HCV cure rate was 90.3% in facilitated telemedicine compared to 39.4% in offsite referral.

In the proposed project, we seek to establish facilitated telemedicine as a standard of care treatment approach at 3 opioid treatment programs operated by the Catholic Health System.

ELIGIBILITY:
Inclusion Criteria:

* evidence of active HCV infection

Exclusion Criteria:

* no evidence of active HCV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals enrolled in the opioid treatment programs of Catholic Health System
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
HCV Treatment Initiation | 1 year
  The time point that HCV treatment is initiated
HCV Sustained Virologic Response | 1 year
  The time point that HCV cure (sustained virologic response) is achieved

CONTACTS AND LOCATIONS:
Overall Officials: Andrew H Talal, MD, MPH, Principal Investigator — University at Buffalo

IPD SHARING:
Plan to Share IPD: Undecided
Data will be de-identified. Available upon reasonable request after publication of study results.

REFERENCES:
- [Background] Talal AH, Markatou M, Liu A, Perumalswami PV, Dinani AM, Tobin JN, Brown LS. Integrated Hepatitis C-Opioid Use Disorder Care Through Facilitated Telemedicine: A Randomized Trial. JAMA. 2024 Apr 23;331(16):1369-1378. doi: 10.1001/jama.2024.2452. PMID 38568601